CLINICAL TRIAL: NCT03701503
Title: The Comparison of PYY, Ghrelin, GLP1, Glucose Level, VAS Level of Satiety, VAS Level of Hunger and Ad Libitum Intake in Obese and Non-Obese Patients After Breakfast With Balanced Macronutrient Composition
Brief Title: The Comparison of PYY, Ghrelin, GLP1, Glucose Level, Level of Satiety, and Ad Libitum Intake in Obese and Non-Obese Patients After Breakfast With Balanced Macronutrient Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: SEAMEO Regional Centre for Food and Nutrition (Other); Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Fiastuti Witjaksono, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GuthormoneOB-NonOB
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: PYY; Ghrelin; Appetite; Gut Hormones; Obesity; VAS of Satiety; VAS of Hunger; GLP - 1
MeSH Terms: conditions — Obesity | interventions — Diet; Adiposity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obese (Experimental): Women age 20-40, with BMI ≥ 25-35 kg/m2 Given a balanced breakfast (Protein 12,4%, carbohydrate 68,2%, fat 22,6%) with calories according to their energy requirement,which is calculated by adding basal metabolic rate (BMR) with additional energy from physical activity.
  Participants' blood was taken before intervention, and 15, 60, 120, and 180 minutes after intervention, then examined in laboratory to measure every outcome. After 4 hours, participants were given ad libitum meal. After the participants done eating, the calorie in meal taken by participants was measured.
  Interventions: Behavioral: Diet with balance composition to know the effect of a meal to gut hormones in obese and non obese women
- Non Obese (Active Comparator): Women age 20-40, with BMI 18,5-23 kg/m2 Given a balanced breakfast (Protein 12,4%, carbohydrate 68,2%, fat 22,6%) with calories according to their energy requirement,which is calculated by adding basal metabolic rate (BMR) with additional energy from physical activity.
  Participants' blood was taken before intervention, and 15, 60, 120, and 180 minutes after intervention, then examined in laboratory to measure every outcome. After 4 hours, participants were given ad libitum meal. After the participants done eating, the calorie in meal taken by participants was measured.
  Interventions: Behavioral: Diet with balance composition to know the effect of a meal to gut hormones in obese and non obese women

INTERVENTIONS:
Behavioral: Diet with balance composition to know the effect of a meal to gut hormones in obese and non obese women

SUMMARY:
Obesity can occur due to an imbalance of energy. This energy balance is greatly influenced by hunger and satiety. Obese person cannot resist hunger, while non obese can control hunger. Gut hormones, such as PYY and ghrelin, are associated with appetite and satiety control. This study's objective is to compare the effect of breakfast with balance composition on gut hormones, glucose and ad libitum intake four hours after breakfast between obese and non obese..

The research methodology was used a clinical trial with 18 obese women and 22 non obese women participants. Subjects were given a balance breakfast (protein 12,4%, carbohydrate 68,2%, fat 22,6%). Gut hormones (PYY, Ghrelin, GLP -1) level , Glucose level and satiety level were measured at 0, 15, 60, 120, and 180 minutes after breakfast. Ad libitum meal was given four hours after breakfast and measured after.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 - 30 (for obese am)
* BMI 18,5 - 23 (for NON- obese am)
* with stable body weight within the last 6 months (body weight change less than 4 kg)
* normal blood glucose level.

Exclusion Criteria:

* Patients who never had breakfast
* patients in weight loss program
* patients consuming lipid-absorption inhibitor or appetite-suppressing drugs
* patients that have had gastrointestinal tract resection.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Ghrelin levels at 0 minute | baseline
  analyzed by ELISA, directly taken after having the breakfast with balance composition in both of the study arm.
Ghrelin levels at 15 minute | 15 minutes
  analyzed by ELISA, taken 15 minutes after having the breakfast with balance composition in both of the study arm.
Ghrelin levels at 60 minute | 60 minutes
  analyzed by ELISA, taken 60 minutes after having the breakfast with balance composition in both of the study arm.
Ghrelin levels at 120 minute | 120 minutes
  analyzed by ELISA, taken 120 minutes after having the breakfast with balance composition in both of the study arm
Ghrelin levels at 180 minute | 180 minutes
  analyzed by ELISA, taken 180 minutes after having the breakfast with balance composition in both of the study arm
PYY levels at 0 minute | baseline
  analyzed by Radioimmunoassay, directly taken after having the breakfast with balance composition in both of the study arm
PYY levels at 15 minute | 15 minutes
  analyzed by Radioimmunoassay, taken 15 minutes after having the breakfast with balance composition in both of the study arm
PYY levels at 60 minute | 60 minutes
  analyzed by Radioimmunoassay, taken 60 minutes after having the breakfast with balance composition in both of the study arm
PYY levels at 120 minute | 120 minutes
  analyzed by Radioimmunoassay, taken 120 minutes after having the breakfast with balance composition in both of the study arm
PYY levels at 180 minute | 180 minutes
  analyzed by Radioimmunoassay, taken 180 minutes after having the breakfast with balance composition in both of the study arm
GLP-1 levels at 0 minute | baseline
  analyzed by ELISA, directly taken after having the breakfast with balance composition in both of the study arm
GLP-1 levels at 15 minute | 15 minutes
  analyzed by ELISA, taken 15 minutes after having the breakfast with balance composition in both of the study arm
GLP-1 levels at 60 minute | 60 minutes
  analyzed by ELISA, taken 60 minutes after having the breakfast with balance composition in both of the study arm
GLP-1 levels at 120 minute | 120 minutes
  analyzed by ELISA, taken 120 minutes after having the breakfast with balance composition in both of the study arm
GLP-1 levels at 180 minute | 180 minutes
  analyzed by ELISA, taken 180 minutes after having the breakfast with balance composition in both of the study arm
Glucose levels at 0 minute | baseline
  analyzed by standard random glucose level from venous blood, directly taken after having the breakfast with balanced composition in both of the study arm
Glucose levels at 15 minute | 15 minutes
  analyzed by standard random glucose level from venous blood, taken 15 minutes after having the breakfast with balanced composition in both of the study arm
Glucose levels at 60 minute | 60 minutes
  analyzed by standard random glucose level from venous blood, taken 60 minutes after having the breakfast with balanced composition in both of the study arm
Glucose levels at 120 minute | 120 minutes
  analyzed by standard random glucose level from venous blood, taken 120 minutes after having the breakfast with balanced composition in both of the study arm
Glucose levels at 180 minute | 180 minutes
  analyzed by standard random glucose level from venous blood, taken 180 minutes after having the breakfast with balanced composition in both of the study arm
Ad Libitum intake | 4 hours
  Mean Ad Libitum intake (calories) in subjects four hours after breakfast with balance composition in both of the study arm
VAS for hunger at 0 minutes | baseline
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), directly taken after having the breakfast with balance composition in both of the study arm
VAS for hunger at 15 minutes | 15 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 15 minutes after having the breakfast with balance composition in both of the study arm
VAS for hunger at 60 minutes | 60 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 60 minutes after having the breakfast with balance composition in both of the study arm
VAS for hunger at 120 minutes | 120 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 120 minutes after having the breakfast with balance composition in both of the study arm
VAS for hunger at 180 minutes | 180 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 180 minutes after having the breakfast with balance composition in both of the study arm
VAS for satiety at 0 minutes | baseline
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), directly taken after having the breakfast with balance composition in both of the study arm
VAS for satiety at 15 minutes | 15 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 15 minutes after having the breakfast with balance composition in both of the study arm
VAS for satiety at 60 minutes | 60 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 60 minutes after having the breakfast with balance composition in both of the study arm
VAS for satiety at 120 minutes | 120 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 120 minutes after having the breakfast with balance composition in both of the study arm
VAS for satiety at 180 minutes | 180 minutes
  Visual Analog Scale, a scale in the form of an empty straight line with no values but only several level point (ex: if the line is 10cm, then each cm represent 1 level). Extreme choices are both ends of the straight line. The minimum value is at the left end and the maximum value is at the right end. The subject must make a choice between the two ends of the line by giving an X mark (ex : if the subject feels less hunger, then the subject should mark X at the second point from far left), taken 180 minutes after having the breakfast with balance composition in both of the study arm

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Nutrition, Faculty of Medicine Universitas Indonesia, Jakarta, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: No